CLINICAL TRIAL: NCT01231061
Title: Randomized Phase II Study of Image-Guided Radiosurgery / SBRT for Localized Spine Metastasis
Brief Title: Spinal met_radiosurgery/SBRT Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYM008
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Spine Metastasis
Keywords: spine metastasis; SBRT; Radiosurgery
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: SBRT (Experimental)
  Interventions: Radiation: SBRT
- Arm B: Radiosurgery (Experimental)
  Interventions: Radiation: Radiosurgery

INTERVENTIONS:
Radiation: SBRT — •24 Gy in 3 fractions to cover at least 90% of the defined target volume
  Arms: Arm A: SBRT
Radiation: Radiosurgery — 16 Gy in 1 fraction to cover at least 90% of the defined target volume
  Arms: Arm B: Radiosurgery

SUMMARY:
Demonstrate the technical feasibility of treating spine metastases with image-guided radiosurgery/SBRT

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have localized spine metastasis from the C1 to L5 levels by a screening imaging study (bone scan, PET, CT, or MRI). A solitary spine metastasis; two separate spine levels; or up to 3 separate sites are permitted. Each of the separate sites may have a maximal involvement of 2 contiguous vertebral bodies. A paraspinal mass ≤ 5 cm is allowed.
2. Zubrod Performance Status 0-2;
3. Age ≥ 18;
4. History/physical examination within 2 weeks prior to registration;
5. No pregnancy for women of childbearing potential;
6. MRI of the involved spine within 4 weeks prior to registration to determine the extent of the spine involvement. MRI is required as it is superior to a CT scan in delineating the spinal cord as well as identifying an epidural or paraspinal soft tissue component. If possible, an MRI with thin slice thickness (<1mm) with 3D reconstruction quality would be most preferable for treatment planning purpose.
7. Numerical Rating Pain Scale within 1 week prior to registration. The patient must have a score on the Scale of ≥ 4 for at least one of the planned sites for spine radiosurgery. Patients taking medication for pain at the time of registration are eligible.
8. Neurological examination within 1 week prior to registration to rule out rapid neurologic decline; see Appendix IV for the standardized neurological examination. Patients with mild to moderate neurological signs are eligible. These neurological signs include radiculopathy, dermatomal sensory change, and muscle strength of involved extremity 4/5 (lower extremity for ambulation or upper extremity for raising arms and/or arm function).
9. Patients with epidural compression are eligible provided that there is no significant displacement or compression on the spinal cord itself.
10. Patients with a paraspinal mass ≤ 5 cm in the greatest dimension and that is contiguous with spine metastasis are eligible.
11. Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Histologies of myeloma or lymphoma.
2. Patients with any spine metastasis with a rating of < 4 on the Numerical Rating Pain Scale.
3. Non-ambulatory patients.
4. Spine instability due to a compression fracture.
5. > 50% loss of vertebral body height.
6. Significant spinal cord compression or displacement.
7. Patients with rapid neurologic decline.
8. Bony retropulsion causing neurologic abnormality.
9. Prior radiation to the index spine.
10. Patients for whom an MRI of the spine is medically contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain control at 3 months post-treatment | 4 years

SECONDARY OUTCOMES:
Determine the time of onset of pain response of the responders at the treated site(s) using radiosurgery/SBRT | 4 years
Determine the duration of pain response at the treated site(s) using radiosurgery/SBRT | 4 years
Study the adverse events of radiosurgery/SBRT according to the criteria in the CTEP Active Version of the CTCAE | 4 years
Evaluate the radiological response of image-guided radiosurgery/SBRT by RECIST MRI | 4 years
2-year Tumor Control Rate | 4 years
Overall Survival | 4 years
Quality of life assessment | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael KM KAM, FRCP, Principal Investigator — Department of Clinical Oncology, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong